CLINICAL TRIAL: NCT07376642
Title: A Phase I/IIa, Open-label, Single-center, Dose-escalation and Dose-expansion Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of IMV101 as a Single Agent in Subjects With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Immunofoco Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMV101-CT01
Record Dates: First submitted 2025-12-29; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: This Phase I/IIa study is an open-label, single-center trial incorporating dose-escalation and dose-expansion cohorts to assess the safety, tolerability, and preliminary antitumor efficacy of IMV101 in subjects with relapsed or refractory B-cell non-Hodgkin lymphoma-including but not limited to diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), primary mediastinal large B-cell lymphoma (PMBCL), and high-grade B-cell lymphoma (HGBCL)-as well as mantle cell lymphoma (MCL).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IMV101 treatment group (Experimental): IMV101 single infusion
  Interventions: Drug: IMV101 treatment

INTERVENTIONS:
Drug: IMV101 treatment — IMV101 Dose Escalation Scheme: Dose Level DL-1，Dose 1e7、Dose Level DL1，Dose 3e7、Dose Level DL2 Dose 1e8、Dose Level DL3 Dose 3e8、Dose Level DL4 Dose 1e9；Accelerated Titration: The 3×10⁷ TU/subject dose cohort will enroll one subject. If this subject experiences a Grade ≥2 adverse event related to IMV101, the cohort will transition to the standard "3+3" design by enrolling two additional subjects for safety and tolerability assessment.

SUMMARY:
A phase I/IIa, open-label, single-center, dose-escalation and dose-expansion study to evaluate the safety, tolerability, and preliminary efficacy of IMV101 as a single agent in subjects with relapsed/refractory B-cell non-Hodgkin Phase I:To observe and evaluate the safety and tolerability of IMV101 in subjects with relapsed/refractory B-cell non-Hodgkin lymphoma.

Phase IIa:To determine the Recommended Phase II Dose (RP2D) based on integrated safety and efficacy data following IMV101 treatment.

To evaluate the preliminary antitumor efficacy of IMV101. Secondary Study Objectives:To evaluate other safety parameters following IMV101 treatment.

To evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) profiles following administration of IMV101.

Exploratory Objective:To evaluate biomarkers change pre- and post-IMV101 administration and their correlation with efficacy and safety.

To perform long-term follow-up for immunogenicity analysis, viral shedding studies, tumor multi-omics research, lentiviral integration sites, and replication-competent lentivirus (RCL), among others.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older, any sex.
2. Previously histologically or cytologically confirmed relapsed/refractory B-cell non-Hodgkin's lymphoma, including the following WHO-defined types: diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), primary mediastinal large B-cell lymphoma (PMBCL), high-grade B-cell lymphoma (HGBCL), and mantle cell lymphoma (MCL), among others.
3. CD19 positivity confirmed by pathology or flow cytometry analysis (subjects with prior exposure to CD19-targeted therapies must undergo repeat biopsy prior to enrollment to reconfirm CD19-positive status).
4. Relapsed/refractory B-cell non-Hodgkin lymphoma meeting at least one of the following criteria:

   1. Disease progression after at least two prior lines of systemic therapy (including relapse, treatment failure, or disease progression), with documented prior exposure to both an anti-CD20 monoclonal antibody (unless CD20-negative) and an anthracycline-based chemotherapy regimen.
   2. Relapsed disease following autologous hematopoietic stem cell transplantation; or relapse occurring ≥2 years after allogeneic hematopoietic stem cell transplantation, in the absence of ongoing immunosuppressive therapy.
   3. Primary refractory disease, defined as stable disease or disease progression as best response after at least two cycles of initial anti-CD20-based immunochemotherapy.

      5． According to the Lugano lymphoma response criteria (Cheson et al, 2014), at least one measurable lesion must be present, meeting one of the following conditions:

   <!-- -->

   1. A nodal lesion with a long axis >15 mm (short axis may be used if measurable).
   2. An extranodal lesion with both long and short axes >10 mm. Lesions previously irradiated will only be considered measurable if documented progression has occurred after radiation therapy.

      6． Life expectancy ≥ 12 weeks. 7． ECOG performance status score of 0 or 1. 8． Subjects must have adequate organ and marrow function. Laboratory screening must meet all of the following criteria, with all values falling within the specified ranges without ongoing supportive care. If any laboratory result is outside these limits, one repeat test is permitted within one week. If the repeat result still does not meet the criteria, the subject fails screening and is ineligible for enrollment:

   <!-- -->

   1. Hematological criteria (in the absence of intensive transfusion [≥2 times within 1 week], platelet administration, or growth factor support [with the exception of recombinant erythropoietin] within 7 days prior to testing).
   2. Hepatic Function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be ≤2.5×ULN, and total bilirubin ≤2×ULN (except in subjects with Gilbert's syndrome); for those with documented hepatic involvement by lymphoma, ALT and AST must be <5×ULN.
   3. Renal Function: Serum creatinine ≤1.5×ULN; if serum creatinine exceeds this threshold, creatinine clearance must be >50 mL/min (calculated using the Cockcroft-Gault formula). Urine protein dipstick must be ≤1+; if dipstick result is ≥2+, 24-hour urine protein quantification is required (acceptable if <1 g/24h).

      9． All toxicities from prior anticancer therapy must have resolved to Grade 0-1 (per NCI CTCAE v5.0) or to a level meeting the study's inclusion/exclusion criteria. Exceptions include alopecia, vitiligo, and other toxicities considered by the investigator to pose no safety risk to the subject.

      10．Reproductive Status: Females of childbearing potential or male subjects with female partners of childbearing potential must be willing to use highly effective medically approved contraception from the time of informed consent until 12 months after IMV101 administration. Acceptable methods include intrauterine devices or condoms (childbearing potential includes premenopausal women and women within 24 months of menopause).

      11． Subjects must provide signed and dated written informed consent. 12．Subjects must demonstrate willingness and ability to comply with the prescribed treatment plan, laboratory tests, follow-up visits, and other study requirements.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Subjects with active central nervous system (CNS) involvement or intestinal parenchymal involvement by B-cell non-Hodgkin lymphoma.
3. Presence of lymphoma cells in cerebrospinal fluid (CSF), brain metastases, or a history of CNS lymphoma, primary CNS lymphoma, or previously detected lymphoma cells in CSF or brain metastases.
4. Subjects with lymphoma infiltration of the atria or ventricles.
5. Subjects who have received or require any of the following treatments/therapies:

   1. Acute or chronic graft-versus-host disease (GVHD) requiring systemic treatment within 4 weeks prior to enrollment.
   2. Requiring immunosuppressive treatment during the study period due to autoimmune diseases (including but not limited to Crohn's disease, rheumatoid arthritis, psoriasis, systemic lupus erythematosus, or asthma requiring bronchodilator intervention), immunodeficiency, or other medical conditions. Exceptions include type 1 diabetes; dermatological conditions not requiring systemic therapy (e.g., vitiligo, psoriasis); alopecia; hypothyroidism managed with hormone replacement therapy only; childhood asthma that has completely resolved with no intervention required in adulthood; or other conditions not expected to recur in the absence of an external trigger.
   3. Received autologous stem cell transplantation (ASCT) within 12 weeks prior to enrollment, or any prior allogeneic hematopoietic stem cell transplantation (allo-HSCT).
   4. Administration of live attenuated vaccines within 4 weeks before the planned IMV101 administration or planned receipt of such vaccines during the 12-week study period.
   5. Systemic corticosteroid use at a dose exceeding 15 mg/day prednisone equivalent for more than 3 days within 2 weeks prior to IMV101 administration, with the exception of inhaled corticosteroids.
   6. Any comorbidities that, in the Investigator's judgment, are expected to require systemic corticosteroid therapy (except for physiological replacement therapy with ≤12 mg/m²/day hydrocortisone or equivalent) or other immunosuppressive agents (excluding topical therapy) within 12 weeks after IMV101 administration;
   7. Participation in another interventional clinical trial with receipt of any investigational product within 1 month prior to the planned administration of the study drug.
   8. Prior to IMV101 administration, subjects who have received any of the following antineoplastic therapies: chemotherapy, targeted therapy, biologic therapy, endocrine therapy, or immunotherapy, where the last dose was administered within 28 days or 5 half-lives (whichever is shorter) before the first IMV101 dose in this study; or have received traditional Chinese medicine with approved antineoplastic indications within 2 weeks prior to IMV101 administration.
   9. Major surgery within 2 weeks prior to enrollment in this study, or planned surgery during the waiting period for IMV101 administration or within 12 weeks after treatment (excluding scheduled procedures under local anesthesia).
6. Subjects with a history of concurrent or previous other malignancies are excluded, except for the following conditions:

   1. Adequately treated basal cell or squamous cell carcinoma (requiring sufficient wound healing prior to enrollment);
   2. Carcinoma in situ of the cervix or breast, treated with curative intent and without evidence of recurrence for at least 3 years prior to the study;
   3. Primary tumor that has been completely resected and in complete remission for ≥5 years.
7. Seropositivity for human immunodeficiency virus (HIV); active hepatitis B virus (HBV) infection (HBV-DNA >10³IU/mL); acute or chronic active hepatitis C (anti-HCV positive); confirmed syphilis seropositivity; active Epstein-Barr virus (EBV) infection (IgM-positive); active cytomegalovirus (CMV) infection (IgM-positive); or SARS-CoV-2 infection confirmed by nucleic acid or antigen testing without documented resolution to negative within 7 days.
8. Active or clinically uncontrolled severe infection; or subjects with bacterial, fungal, or viral infections requiring intravenous antibiotic therapy who, in the judgment of the Investigator, are unsuitable for study participation; or subjects on prophylactic antibiotic therapy who, in the judgment of the Investigator, may continue in the study.
9. Uncontrolled pleural effusion, pericardial effusion, or ascites present prior to participation in this study.
10. Oxygen saturation≤95% while on nasal cannula oxygen.
11. Presence of other significant pulmonary diseases that may limit participation in this study, such as pulmonary embolism, chronic obstructive pulmonary disease, symptomatic or poorly controlled interstitial lung disease, or clinically significant abnormalities in pulmonary function tests.
12. Known history or current presence of hepatic encephalopathy requiring treatment; subjects with current or historical central nervous system disorders, including but not limited to seizures, cerebral ischemia/hemorrhage, dementia, cerebellar diseases, or any autoimmune disease involving the CNS.
13. Poorly controlled hypertension as determined by the Investigator (defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure >100 mmHg despite standardized antihypertensive therapy); or hypotension requiring vasopressors; or poorly controlled diabetes despite standard treatment (fasting blood glucose ≥10.2 mmol/L).
14. History of any of the following cardiac symptoms or diseases within 6 months prior to IMV101 administration:

    1. Left ventricular ejection fraction (LVEF) < 50%;
    2. Myocardial infarction within 1 year; or unstable angina; or history of percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG); or use of a cardiac pacemaker;
    3. QTc interval > 450 ms (male) or > 470 ms (female) on resting electrocardiogram (ECG)
    4. Clinically significant abnormalities on resting ECG (e.g., abnormalities in heart rate, conduction, or morphology) or complete left bundle branch block, third-degree atrioventricular block, or PR interval > 250 ms.
15. History of other severe allergic reactions, such as anaphylaxis.
16. Subjects with severe psychiatric disorders.
17. Subjects with newly developed arrhythmias, including but not limited to those not adequately controlled by antiarrhythmic medication.
18. History of solid organ transplantation.
19. Subjects who, in the opinion of the Investigator, are unable or unwilling to comply with the requirements of the study protocol.
20. Presence of any other concurrent severe and/or uncontrolled medical condition that, based on the Investigator's judgment, renders the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
DLTs/RP2D/Efficacy endpoint | For dose-limiting toxicity (DLT) assessment: From study drug administration through 28 days after dosing.The Recommended Phase 2 Dose (RP2D) will be evaluated and confirmed by the Study Monitoring Committee (SMC) after discussion.
  To observe the incidence of dose-limiting toxicities (DLTs) within 28 days following IMV101 administration.To determine the Recommended Phase II Dose (RP2D) of IMV101.Efficacy endpoints: Time to response (TTR), objective response rate (ORR), disease control rate (DCR), duration of response (DOR), progression-free survival (PFS), and overall survival (OS). Objective response rate includes stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR), assessed according to the Lugano 2014 classification for lymphoma efficacy assessment (Cheson, 2014).

SECONDARY OUTCOMES:
Treatment-related adverse events (TRAEs) | From first dose of IMV101 until disease progression, initiation of other anti-cancer therapy, or death (whichever occurs first); maximum 15 years of assessment.
  Assessment of the incidence and severity of treatment-related adverse events (TRAEs) will be conducted according to the NCI CTCAE version 5.0, with the exception of CRS and ICANS, which will be graded per the 2019 ASTCT consensus criteria.
Assessment of pharmacokinetic (about Cmax) | From first dose of IMV101 until disease progression, initiation of other anti-cancer therapy, or death (whichever occurs first);maximum 96 weeks of assessment for PK and PD
  The maximum concentration of CAR-T cells in peripheral blood after administration (Cmax)
Assessment of pharmacokinetic (about Tmax) | From first dose of IMV101 until disease progression, initiation of other anti-cancer therapy, or death (whichever occurs first);maximum 96 weeks of assessment for PK and PD
  The time to reach the maximum concentration (Tmax)
Assessment of pharmacokinetic (about AUC0-28d) | From first dose of IMV101 to 28 days after IMV101 administration
  The area under the CAR-T concentration versus time curve (AUC) for 28 days after IMV101 administration
Assessment of pharmacokinetic (about AUC0-90d) | From first dose of IMV101 to 90 days after IMV101 administration
  The area under the CAR-T concentration versus time curve (AUC) for 90 days after IMV101 administration
Evaluation of Pharmacodynamic | From first dose of IMV101 until disease progression, initiation of other anti-cancer therapy, or death (whichever occurs first); maximum 15 years of assessment.
  Concentration levels of CAR-T related serum cytokines such as CRP, IL-6, INF-γ at each time point

OTHER OUTCOMES:
To evaluate the immunogenicity of IMV101 injection | From first dose of IMV101 until disease progression, initiation of other anti-cancer therapy, or death (whichever occurs first); maximum 15 years of assessment.
  The positive rate of human anti-CAR antibody at each time point
RCL testing | From first dose of IMV101 until disease progression, initiation of other anti-cancer therapy, or death (whichever occurs first); maximum 15 years of assessment.
  To detect the presence of replication-competent lentivirus (RCL) in peripheral blood.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing GoBroad Boren Hospital, Beijing, Beijing Municipality
  - Zhengzhou Yihe Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No